CLINICAL TRIAL: NCT00050791
Title: Leptin Treatment for Prevention of the Metabolic and Endocrine Sequelae of a Decreased Caloric Intake: Studies of Patients on a Very Low Calorie Diet
Brief Title: Effects of Leptin Treatment on Weight Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Weill Medical College of Cornell University (Other); St. Luke's-Roosevelt Hospital Center (Other); Columbia University (Other)
Responsible Party: Jeffrey M. Friedman,, MD, PhD, Rockefeller University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JFN 0357
Record Dates: First submitted 2002-12-19; First posted 2002-12-23 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Obesity
Keywords: Obesity; Weightloss; Leptin; Diet; Reducing; Overweight; Fat
MeSH Terms: conditions — Obesity; Weight Loss; Overweight; Platelet Glycoprotein IV Deficiency | interventions — Leptin; recombinant methionyl human leptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VLCD and leptin (Experimental): Very low calorie diet formula providing 800 calories per day and leptin treatment.
  Interventions: Drug: Leptin
- placebo (Active Comparator): Very low calorie diet and placebo treatment
  Interventions: Behavioral: Very Low Calorie Diet

INTERVENTIONS:
Drug: Leptin — Leptin is an adipocyte hormone that functions as an afferent signal in a feedback loop regulating body weight
  Other Names: A-100; Recombinant-methionyl Human Leptin (r-metHuLeptin)
  Arms: VLCD and leptin
Behavioral: Very Low Calorie Diet — placebo injections
  Arms: placebo

SUMMARY:
This is a double blind placebo controlled clinical study designed to determine the effects of leptin on the changes that occur in the body during weight loss achieved by a very low calorie diet.

DETAILED DESCRIPTION:
Leptin is a hormone that is produced by the fat tissue and acts on the brain. Leptin plays a key role in regulating energy balance and body weight in animals and in humans.

When a person loses weight, leptin concentration in the blood is reduced. Reduction in blood leptin levels has been found to be related to a decreased metabolic rate (the rate in which the body burns its calories), an increased appetite, and to many other physiological and hormonal changes that may lead to failure in dieting.

This study is aimed to test if maintaining leptin in the pre-diet level range will ameliorate the changes that occur in the body during weight loss. If these changes are reduced, the process of weight loss could be easier and faster when adhering to a low calorie diet.

In this study, leptin or placebo is administered by an injection under the skin, in a way that is similar to injections of insulin to diabetic patients. 50% of the subjects participating in the study are treated by leptin and 50% are treated by placebo. Blood leptin levels are maintained in the pre-diet range in leptin treated subjects by leptin treatment. Subjects treated by placebo will also lose weight if they adhere to the liquid diet provided by the Rockefeller University Bio-nutrition Department. The investigators and the participants don't know if leptin or placebo are used since this is a double blind study.

To participate in this study, subjects have to stay at the Rockefeller University Hospital as inpatients for about two months and continue the study as outpatients for 4 more months. During the outpatient period, subjects have to attend a clinic visit once a week. During the first 3 weeks of the study, subjects are introduced to a weight stabilization liquid diet. During this time, the initial weight is maintained and baseline study tests are performed. When testing is completed, a very low calorie liquid diet and leptin or placebo administration are initiated. Weight is monitored until 10% weight loss is achieved. At this time, a second testing period is performed in an inpatient setting. When testing is completed, weight loss and leptin or placebo treatment continue at home in an outpatient setting until 20% weight loss is achieved. When this period is completed, a third testing period is performed in an inpatient setting. The last month of the study is dedicated to a transition from the liquid diet to solid food, and to weight maintenance education provided by the hospital staff in an outpatient setting. A solid food weight maintenance diet is provided to participants during this period. At the end of this period, two days of testing are performed and leptin/placebo administration is discontinued.

Study testing periods are performed over 12 days in an inpatient setting and include a variety of blood draws, urine collection, and metabolic and behavioral tests that are known to be affected by weight loss.

ELIGIBILITY:
Inclusion Criteria:

(1) adult females, age 25-45 with BMI 29-45, and no other acute or chronic illnesses. Pregnant women will not be permitted to participate in the study.

Exclusion Criteria:

1. Chronic illnesses other the than mild forms illnesses related to obesity (hypertension, hyperlipidemia etc) that do not require medical treatment
2. Diabetes Mellitus
3. Chronic drug treatment for any medical conditions
4. Inability to give informed consent
5. Inability to give contact information (for outpatient follow up) including permanent residence, provide evidence of a stable living environment for the study period.
6. Active weight reduction of more than 7 pounds in the last 3 months
7. Weight at screening more than 6% lower than the maximal life time weight.
8. History of bleeding or blood clotting disorders.
9. Changes in smoking habits for the last 3 months.
10. Pregnancy or breast feeding in women.
11. Allergic reaction to local anesthetics
12. History of anaphylaxis or anaphylactoid-like reactions
13. Tendency to form scars (keloids) easily
14. Subjects with known hypersensitivity to E Coli-derived proteins or any other component of the A-100 preparation.
15. Irregular menses
16. HIV and hepatitis B or C positive subjects.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2001-03; Primary Completion 2006-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
energy expenditure after 10% and 20% weight loss, achieved by a VLCD with or without A-100 treatment | Testing period 2,3 and 4 after 10% and 20% weight loss

SECONDARY OUTCOMES:
endocrine and behavioral parameters | testing period 2, 3 and 4. After 10% and 20% weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Friedman, MD, PHD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States